CLINICAL TRIAL: NCT00161135
Title: Magnetic Resonance Imaging in Children and Adolescents With Autism and Multiple Complex Developmental Disorders
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Other Study IDs: WOM 98/261
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Autism; Developmental Disabilities
Keywords: MRI; PDD-NOS, MCDD
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the overlap and differences between autism and MCDD as neuropsychiatric childhood disorders. MRI scans are acquired from subjects with autism, subjects with a diagnosis of MCDD and typically developing controls. Volumetric measure of various brain regions are compared between groups. We hypothesize that subjects with autism will have larger brains than controls, whereas subjects with MCDD will have smaller brains.

DETAILED DESCRIPTION:
Autism and Childhood-onset Schizophrenia have been clearly defined as neuropsychiatric disorders since the studies of Kolvin and Rutter. In the early seventies the discussion on a possible overlap between the two types of disorders vanished, but nowadays this issue revives. Amongst all the advances of the DSM diagnostic criteria, the omission of developmental information appears to be a disadvantage. The Pervasive Developmental Spectrum is a broad spectrum, that with exceptions for Autism and some other characteristic disorders, to a large extent consists of an ill-defined restcategory. Most patients actually belong to this last category , the so-called PDD-NOS group. In recent years more has been published about the subgroups within this large group. One of these subgroups, the Multiple Complex Developmental Disorder (MCDD), appears to be a well defined category of patients whose validity has been confirmed by research. In adulthood, a large percentage of this MCDD group seems to develop Schizophrenia or a Schizophrenia related disorder. This again does arise the question of a possible overlap. This discussion is even emphasized by reports notably on -mostly retrospective- studies of premorbid autistic features in patients with Schizophrenia.

In the present day studies on neurodevelopmental psychiatric disorders, there is a search for biological markers or discriminating factors. One of the applied methods is structural imaging. Question marks can be placed on the differing study set-ups and protocols which seriously hinder their inter alia comparison. However one can still conclude that the results of studies on subjects with Autism and Childhood-onset Schizophrenia reveal major differences. However, structural abnormalities do not tell anything about possible functional abnormalities. But detecting structural abnormalities can be helpful in forming hypothesis about the origin of these neurodevelopmental disorders.

In this study brain structures will be measured by magnetic resonance imaging. Structural deviances will be interpreted as a reflection of functional abnormalities. It is hypothesized that the abnormalities on structural imaging in MCDD patients will more resemble the abnormalities found in the literature for (Childhood-onset) Schizophrenia instead of the deviances revealed in subjects with Autism.

In this study patients with Autism and MCDD will be divided in two groups: before and after puberty. Each group will behold 15-40 subjects. They each will be compared with two groups of 20-25 age, sex and IQ matched controls. They will participate in carrying out a MRI scan, filling in some questionnaires and if necessary an IQ test and a general physical examination.The MRI scans will be measured, and compared with each other in order to find 'disorder-specific' abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism according to ADI-interview or diagnosis of MCDD according to the MCDD-checklist or no psychiatric diagnosis (controls)

Exclusion Criteria:

* Some medical and neurological diseases (if there are influences on the brain structures)
* Alcohol or drug abuse
* IQ < 70
* Focal abnormalities on the MRI scan

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Bertine E Lahuis, M.D., Principal Investigator — Rudolf Magnus Institute of Neuroscience, University Medical Center Utrecht; Sarah Durston, Ph.D., Study Director — Rudolf Magnust Institute of Neuroscience, UMC Utrecht; Herman van Engeland, M.D. Ph.D., Study Chair — Rudolf Magnus Institute of Neuroscience, UMC Utrecht
Locations (1):
- Dept. of Child and Adolescent Psychiatry, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Palmen SJ, Hulshoff Pol HE, Kemner C, Schnack HG, Durston S, Lahuis BE, Kahn RS, Van Engeland H. Increased gray-matter volume in medication-naive high-functioning children with autism spectrum disorder. Psychol Med. 2005 Apr;35(4):561-70. doi: 10.1017/s0033291704003496. PMID 15856726
- [Result] Palmen SJ, Hulshoff Pol HE, Kemner C, Schnack HG, Janssen J, Kahn RS, van Engeland H. Larger brains in medication naive high-functioning subjects with pervasive developmental disorder. J Autism Dev Disord. 2004 Dec;34(6):603-13. doi: 10.1007/s10803-004-5282-2. PMID 15679181